CLINICAL TRIAL: NCT04847700
Title: Minimally Invasive Vestibular Neurectomy Versus Tenotomy of the Stapedius and Tensor Tympani Muscles in the Management of Patients With Unilateral Meniere's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha A.Elkholy, Principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.21.02.418.R1
Record Dates: First submitted 2021-03-26; First posted 2021-04-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Ménière
MeSH Terms: conditions — Meniere Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive vestibular neurectomy (Active Comparator)
  Interventions: Procedure: Surgical treatment
- Tenotomy of the stapedius and tensor tympani muscles (Active Comparator)
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Endoscopic retrosigmoid minimally invasive vestibular neurectomy
  Arms: Minimally invasive vestibular neurectomy
Procedure: Surgical treatment — Endoscopic tenotomy of middle ear muscles
  Arms: Tenotomy of the stapedius and tensor tympani muscles

SUMMARY:
The distinctive symptoms of Meniere's disease (MD) include recurrent vertigo spells, fluctuating hearing loss, aural fullness and tinnitus. Conservative treatment in MD comprises lifestyle modifications, such as low-sodium diet, avoidance of caffeine, alcohol and stress, in addition to medication such as diuretics and betahistine. When conservative treatment fails, surgical management is attempted. Surgical interventions comprise transtympanic steroids or gentamicin, endolymphatic sac surgery (ES), ventilation tube placement, vestibular neurectomy, and labyrinthectomy. Recently, Loader et al. have presented encouraging results of the effectiveness of tenotomy of the stapedius and tensor tympani muscles (TSTM) in the management of patients with definite MD. Also, satisfactory results were obtained with endoscopic assisted minimally invasive vestibular neurectomy (MIVN). The aim of this study is to compare the clinical outcomes of MD patients who were submitted to either MIVN or TSTM in our department.

ELIGIBILITY:
Inclusion Criteria:

* unilateral definite Meniere's disease.

Exclusion Criteria:

* other peripheral or central vestibular disorders, bilateral MD and neurologic disorders.
* Previous history of chronic otitis media or middle ear surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
dizziness handicap inventory (DHI) | 6 months after surgery
  contains 25 questions divided into physical, emotional, and functional subgroups. Each question is to be answered using a scale with ''no'' (0 points), ''sometimes'' (2 points), or ''yes'' (4 points). The total score ranges from zero (no incapacity) to 100 (severe incapacity).

CONTACTS AND LOCATIONS:
Locations (1):
- ORL-HNS department,Mansoura University Hospital, Faculty of Medicine, Mansoura University, Al Mansurah, ElDakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No